CLINICAL TRIAL: NCT06174584
Title: Comparison of Cow Milk and 15% Hypertonic Saline in the Treatment of Rectal Prolapse in Children
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, Mansoor Ahmed, Principal Investigator, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ShaheedZABMU1234
Record Dates: First submitted 2023-11-28; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Rectal Prolapse
MeSH Terms: conditions — Rectal Prolapse | interventions — Saline Solution, Hypertonic; Milk

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cow Milk (Active Comparator): Cow Milk was injected as sclerosing agent in one group
  Interventions: Other: Cow Milk
- 15% Hypertonic Saline (Active Comparator): Hypertonic Saline 15% used as sclerosing agent in other half.
  Interventions: Drug: Hypertonic saline

INTERVENTIONS:
Drug: Hypertonic saline — Hypertonic saline
  Arms: 15% Hypertonic Saline
Other: Cow Milk — Cow Milk
  Arms: Cow Milk

SUMMARY:
To see the outcome of results of Cow Milk & Hypertonic Saline in the treatment of Rectal Prolapse in Children

DETAILED DESCRIPTION:
Sclerotherapy is the least invasive procedure used in management of grade I/II rectal prolapse, with a success rate of around 80%, and generally considered as the first choice for uncomplicated and recurrent prolapse. Several sclerosing agents such as 15% hypertonic saline, 5% Phenol in almond oil and cow milk have been used and reported in the literature. Present study is designed to determine the efficacy of cow milk and 15% hypertonic saline in the management of children with grade I/II rectal prolapse.

All the details will be entered on the proforma which will include resolvement of rectal prolapse and which agent has adverse effects like recurrence, fecal incontinence and anal stenosis.

ELIGIBILITY:
Inclusion Criteria:

* All children with Grade I and II rectal prolapse
* Age <12 years
* Both genders

Exclusion Criteria:

* Rectal prolapse secondary to causes like ulcerative colitis and crohn's disease
* Past surgical history on the pelvic floor,
* Neurological diseases like rectal polyps, congenital megacolon, Hirschsprung disease, sacrococcygeal teratoma, neural tube defects, cauda equina syndrome
* Where parents are not willing to participate in the study

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
recurrence (as described by parent s during follow up) | 1 year
  Comparison of Cow Milk vs 15% Hypertonic Saline for rectal prolapse
Number of participants with fecal incontinence (as described by parents during follow up) | 1 year
  Comparison of Cow Milk vs 15% Hypertonic Saline for rectal prolapse
Number of participants with anal stenosis (on clinical examination) | 1 year
  Comparison of Cow Milk vs 15% Hypertonic Saline for rectal prolapse

CONTACTS AND LOCATIONS:
Overall Officials: Mansoor Ahmed, MBBS, Principal Investigator — Shaheed Zulfiqar Ali Bhutto Medical University
Locations (1):
- Shaheed Zulfiqar Ali Bhutto Medical University/PIMS, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No
Confidentiality